CLINICAL TRIAL: NCT02832765
Title: Intensity-modulated Radiotherapy With Integrated-boost in Patients With Spinal Bone Metastases
Acronym: IRON-2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRON-2
Record Dates: First submitted 2016-07-12; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Vertebral Bony Metastases
Keywords: Palliative radiotherapy; Bone metastases
MeSH Terms: interventions — Fumigant 93

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Intensity modulated radiotherapy (IMRT) 30Gy in 10 fractions
  Interventions: Radiation: A
- B (Experimental): Intensity modulated radiotherapy (IMRT) 30Gy in 10 fractions with an SIB with 40 Gy in 10 fractions to the metastasis
  Interventions: Radiation: B
- C (Experimental): Intensity modulated radiotherapy (IMRT) 20Gy in 5 fractions
  Interventions: Radiation: C
- D (Experimental): Intensity modulated radiotherapy (IMRT) 20Gy in 5 fractions with an SIB with 30 Gy in 5 fractions to the metastasis
  Interventions: Radiation: D

INTERVENTIONS:
Radiation: A — Intensity modulated radiotherapy (IMRT) 30Gy in 10 fractions of the involved spinal bone metastases
  Arms: A
Radiation: B — Intensity modulated radiotherapy (IMRT) 30Gy in 10 fractions with an SIB with 40 Gy in 10 fractions to the metastasis of the involved spinal bone metastases
  Arms: B
Radiation: C — Intensity modulated radiotherapy (IMRT) 20Gy in 5 fractions of the involved spinal bone metastases
  Arms: C
Radiation: D — Intensity modulated radiotherapy (IMRT) 20Gy in 5 fractions with an SIB with 30 Gy in 5 fractions to the metastasis of the involved spinal bone metastases
  Arms: D

SUMMARY:
The primary goal of the study is to determine the local control-rate after radiotherapy (RT) with and without simultaneous integrated boost (SIB) concepts in patients with bone metastases of the spine. Further study objectives are survival, and clinical parameters such as pain, quality of life (QoL) and fatigue. We expect an improvement in local control and consecutively an increased re-sclerotization of the bone metastasis due to a higher biological dose in the tumor area. Therefore patients could benefit in quality-of-life, pain relief and mobility.

DETAILED DESCRIPTION:
The vertebral column is the main localization of bone metastases and is where they frequently indicate an advanced stage of a malignant primary disease [1, 2]. Two thirds of all patients with tumors are estimated to develop bone metastases in the course of their disease [3]. Spinal bone metastases are of central impact for patients in a palliative setting. The clinical symptoms include pain at rest and under exercise but also impaired activity of daily life, the risk of pathological fractures, and neurological deficits. Local control is the essential factor for stability of the vertebral body of patients with spinal bone metastases. In regard to re-calcification of former osteolytic lesions, palliative radiotherapy (RT) represents an effective treatment option [4]. The most common schedule was specified as 30 Gy in 10 fractions. Stereotactic body radiation therapy (SBRT) using intensity-modulated radiotherapy (IMRT) can be a safe modality for treating spinal metastasis with enhanced targeting accuracy [5]. Secondly, IMRT to the spine was well tolerated (especially in the spinal cord), had no significant late toxicities, and spared other organs at risk simultaneously [6]. The main problem of the standard schedule is the limited dose application to the metastasis due to organ at risk myelon. Therefore, the aims of this study is to apply a high biological dose in the tumor region and to achieve an improved result related to local control for palliative patients with painful spinal bone metastases. Secondly, the aim is to evaluate QoL, fatigue, and survival of three different RT-techniques. To the best of our knowledge, no comparable randomized study has been described in the literature so far.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologically confirmed tumor diagnosis, with secondarily diagnosed solitary/multiple metastatic spinal bone metastases
* Indication for RT of the bone metastasis
* Age: between 18 and 80 years
* Karnofsky performance score ≥ 70
* Signed Declaration of Informed Consent
* Bisphosphonate therapy

Exclusion Criteria:

* Significant neurological or psychiatric disorders, including dementia and epileptic seizures
* Lacking or diminished legal capacity
* foregoing radiotherapy in the planned RT area
* Any medical of psychological condition that the study director considers a preventive factor for the patient's ability to complete the study or to adequately understand the scope of the study and to give his/her consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
local control | 3 months after RT
  local control as bone density is assessed 12 weeks post completion of radiotherapy using follow-up CT scan of the spine

SECONDARY OUTCOMES:
progression-free survival (PFS) | 2 years post completion of radiotherapy
  PFS is assessed 2 years post completion of radiotherapy
pain reduction | end of treatment, 12 and 24 weeks post completion of radiotherapy
  pain is evaluated using the VAS pain scale (0-100 points) at completion and 12/ 24 weeks post completion of radiation
Quality of life | 12 and 24 weeks post completion of therapy
  Quality of life is assessed using the EORTC BM22 questionnaire at 12 and 24 weeks post completion of treatment
Fatigue | 12 and 24 weeks post completion of therapy
  Fatigue is assessed using the EORTC FA13 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, Germany, Heidelberg, Germany, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ryu S, Pugh SL, Gerszten PC, Yin FF, Timmerman RD, Hitchcock YJ, Movsas B, Kanner AA, Berk LB, Followill DS, Kachnic LA. RTOG 0631 phase 2/3 study of image guided stereotactic radiosurgery for localized (1-3) spine metastases: phase 2 results. Pract Radiat Oncol. 2014 Mar-Apr;4(2):76-81. doi: 10.1016/j.prro.2013.05.001. Epub 2013 Jun 4. PMID 24890347
- [Result] Guckenberger M, Sweeney RA, Flickinger JC, Gerszten PC, Kersh R, Sheehan J, Sahgal A. Clinical practice of image-guided spine radiosurgery--results from an international research consortium. Radiat Oncol. 2011 Dec 15;6:172. doi: 10.1186/1748-717X-6-172. PMID 22172095
- [Result] Katsoulakis E, Riaz N, Cox B, Mechalakos J, Zatcky J, Bilsky M, Yamada Y. Delivering a third course of radiation to spine metastases using image-guided, intensity-modulated radiation therapy. J Neurosurg Spine. 2013 Jan;18(1):63-8. doi: 10.3171/2012.9.SPINE12433. Epub 2012 Oct 26. PMID 23101946
- [Result] Chung Y, Yoon HI, Kim JH, Nam KC, Koom WS. Is helical tomotherapy accurate and safe enough for spine stereotactic body radiotherapy? J Cancer Res Clin Oncol. 2013 Feb;139(2):243-8. doi: 10.1007/s00432-012-1321-0. Epub 2012 Oct 2. PMID 23052695
- [Derived] Sprave T, Welte SE, Bruckner T, Forster R, Bostel T, Schlampp I, Nicolay NH, Debus J, Rief H. Intensity-modulated radiotherapy with integrated-boost in patients with bone metastasis of the spine: study protocol for a randomized controlled trial. Trials. 2018 Jan 22;19(1):59. doi: 10.1186/s13063-018-2452-7. PMID 29357902